CLINICAL TRIAL: NCT04144179
Title: Safety and Immunogenicity of Quadrivalent Recombinant Influenza Vaccine Formulations Containing Different H3 Hemagglutinin Antigens in Healthy Adult Subjects 18 to 30 Years of Age
Acronym: FBP00001
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: FBP00001; U1111-1223-4988 (Registry Identifier: ICTRP); FBP00001 (Other: Sanofi Identifier)
Record Dates: First submitted 2019-10-28; First posted 2019-10-30 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Quadrivalent RIV with H3 strain 1 (Experimental): 1 injection of Quadrivalent RIV containing H3 strain 1
  Interventions: Biological: Quadrivalent RIV with H3 strain 1
- Quadrivalent RIV with H3 strain 2 (Experimental): 1 injection of Quadrivalent RIV containing H3 strain 2
  Interventions: Biological: Quadrivalent RIV with H3 strain 2
- Quadrivalent RIV with H3 strain 3 (Experimental): 1 injection of Quadrivalent RIV containing H3 strain 3
  Interventions: Biological: Quadrivalent RIV with H3 strain 3
- Quadrivalent RIV with H3 strain 4 (Experimental): 1 injection of Quadrivalent RIV containing H3 strain 4
  Interventions: Biological: Quadrivalent RIV with H3 strain 4
- Quadrivalent RIV Control (Active Comparator): 1 injection of Quadrivalent RIV containing 2018-19 NH recommended H3 strain
  Interventions: Biological: Quadrivalent RIV with 2018-2019 NH H3 strain

INTERVENTIONS:
Biological: Quadrivalent RIV with H3 strain 1 — Pharmaceutical form: Pre-filled single-dose vial Route of administration: Intramuscular
  Arms: Quadrivalent RIV with H3 strain 1
Biological: Quadrivalent RIV with H3 strain 2 — Pharmaceutical form: Pre-filled single-dose vial Route of administration: Intramuscular
  Arms: Quadrivalent RIV with H3 strain 2
Biological: Quadrivalent RIV with H3 strain 3 — Pharmaceutical form: Pre-filled single-dose vial Route of administration: Intramuscular
  Arms: Quadrivalent RIV with H3 strain 3
Biological: Quadrivalent RIV with H3 strain 4 — Pharmaceutical form: Pre-filled single-dose vial Route of administration: Intramuscular
  Arms: Quadrivalent RIV with H3 strain 4
Biological: Quadrivalent RIV with 2018-2019 NH H3 strain — Pharmaceutical form: Pre-filled single-dose vial Route of administration: Intramuscular
  Arms: Quadrivalent RIV Control

SUMMARY:
The primary objectives of the study are:

* To describe the safety profile of the different quadrivalent recombinant influenza vaccine (RIV) formulations.
* To describe the hemagglutination inhibition (HAI) and seroneutralization (SN) antibody responses against hemagglutinin (HA) (H1, H3, B/Victoria, and B/Yamagata) antigens present in the control vaccine in all groups at all timepoints.

The secondary objectives of the study are:

* To describe antigenic coverage in each group by assessing the HAI and SN antibody responses against a panel of H3 antigens (not present in any of the vaccine formulations).
* To describe HAI and SN antibody responses in each group against each of the H3 antigens.
* To compare the HAI and SN antibody responses for the groups with different H3 antigens to the control group.

DETAILED DESCRIPTION:
Study duration per participant is approximately 90 days.

ELIGIBILITY:
Inclusion criteria :

* Aged 18 to 30 years on the day of inclusion
* Informed consent form has been signed and dated
* Able to attend all scheduled visits and to comply with all study procedures

Exclusion criteria:

* Participant is pregnant, or lactating, or of childbearing potential and not using an effective method of contraception or abstinence from at least 4 weeks prior to vaccination until at least 12 weeks after vaccination. To be considered of non-childbearing potential, a female must be pre-menarche, or post-menopausal for at least 1 year, or surgically sterile
* Participation at the time of study enrollment (or in the 4 weeks preceding the study vaccination) or planned participation during the present study period in another clinical study investigating a vaccine, drug, medical device, or medical procedure
* Receipt of any vaccine in the 4 weeks preceding the study vaccination or planned receipt of any vaccine in the 4 weeks following study vaccination
* Previous vaccination against influenza in the previous influenza season (2018-2019) with any licensed or investigational influenza vaccine
* Previous vaccination against influenza in the 2019-2020 season with any licensed influenza vaccine
* Receipt of immune globulins, blood or blood-derived products in the past 3 months
* Known or suspected congenital or acquired immunodeficiency; or receipt of immunosuppressive therapy, such as anti-cancer chemotherapy or radiation therapy, within the preceding 6 months; or long-term systemic corticosteroid therapy (prednisone or equivalent for more than 2 consecutive weeks within the past 3 months)
* Have known active or recently active (12 months) neoplastic disease or a history of any hematologic malignancy
* History of influenza infection during the 2018-2019 or 2019-2020 influenza season, confirmed by laboratory tests (including rapid tests)
* Self-reported or documented seropositivity for human immunodeficiency virus, hepatitis B, or hepatitis C
* Known systemic hypersensitivity to any of the vaccine components, or history of a life-threatening reaction to the vaccines used in the study or to a vaccine containing any of the same substances
* Thrombocytopenia or bleeding disorder, contraindicating intramuscular vaccination based on Investigator's judgement
* Deprived of freedom by an administrative or court order, or in an emergency setting, or hospitalized involuntarily
* Alcohol abuse or substance abuse that, in the opinion of the investigator, might interfere with the study conduct or completion
* Chronic illness that, in the opinion of the investigator, is at a stage where it might interfere with study conduct or completion or predispose to complications associated with influenza infection
* Have any diagnosis, current or past, of chronic pulmonary diseases including asthma, cystic fibrosis and chronic pulmonary obstructive disease
* Have taken high-dose inhaled corticosteroids within 6 months prior to study vaccination
* Body Mass Index of 40 or higher
* History of cardiac disease such as congenital heart disease, heart failure, coronary artery disease (except isolated hypertension)
* Health care personnel in inpatient and outpatient care settings, medical emergency-response workers, employees of nursing home and long-term care facilities who have contact with patients or residents and students in these professions who will have contact with patients
* Moderate or severe acute illness/infection (according to investigator judgment) on the day of vaccination or febrile illness (temperature ≥ 100.4 F [≥ 38.0 C]). A prospective participant should not be included in the study until the condition has resolved or the febrile event has subsided
* Identified as an Investigator or employee of the Investigator or study center with direct involvement in the proposed study, or identified as an immediate family member (ie, parent, spouse, natural or adopted child) of the Investigator or employee with direct involvement in the proposed study
* Personal or family history of Guillain-Barré syndrome

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2019-11-06 (Actual); Primary Completion 2020-02-24 (Actual); Study Completion 2020-02-24 (Actual)

PRIMARY OUTCOMES:
Number of participants with immediate adverse events | Within 30 minutes after vaccination
  Immediate adverse events are unsolicited systemic adverse events reported in the 30 minutes after vaccination
Number of participants with solicited injection site or systemic reactions | From Day 0 to Day 7
  Solicited injection site reactions: injection site pain, erythema, swelling, induration and bruising; solicited systemic reactions: fever, headache, malaise, and myalgia
Number of participants with unsolicited adverse events | From Day 0 to Day 28
  Unsolicited (spontaneously reported) adverse events not fulfilling criteria for solicited reactions
Number of participants with serious adverse events | From Day 0 to Day 90
  Serious adverse events are collected throughout the study
Number of participants with adverse events of special interest | From Day 0 to Day 90
  Adverse events of special interest are collected throughout the study
HAI antibody titers against HA influenza antigens in quadrivalent RIV control group | From Day 0 to Day 90
  Influenza vaccine antigens are measured by HAI assay
Individual ratio of HAI titers against HA influenza antigens in quadrivalent RIV control group | From Day 0 to Day 90
  Titers ratio are calculated for Day 8/Day 0 and Day 28/Day 0, Day 56/Day 28 and Day 90/Day 28
Number of participants with seroconversion to HA influenza antigens in quadrivalent RIV control group | Day 28
  Seroconversion is defined as HAI antibody titer < 10 [1/dil] at Day 0 and post-injection titer ≥ 40 [1/dil] at Day 28, or titer ≥ 10 [1/dil] at Day 0 and a ≥ 4-fold increase in titer [1/dil] at Day 28
Number of participants with HAI antibody titer ≥ 40 [1/dil] against HA influenza antigens in quadrivalent RIV control group | From Day 0 to Day 90
  Influenza vaccine antigens are measured by HAI assay

SECONDARY OUTCOMES:
2-fold and 4-fold increase in SN antibody titers against HA influenza antigens in quadrivalent RIV control group | From Day 0 to Day 90
HAI and SN antibody titers against influenza H3 antigens | From Day 0 to Day 90
Individual ratio of HAI and SN titers against influenza H3 antigens | From Day 0 to Day 90
  Titers ratio are calculated for Day 8/Day 0 and Day 28/Day 0, Day 56/Day 28 and Day 90/Day 28
Number of participants with seroconversion to influenza H3 antigens | Day 28
  Seroconversion is defined as HAI antibody titer < 10 [1/dil] at Day 0 and post-injection titer ≥ 40 [1/dil] at Day 28, or titer ≥ 10 [1/dil] at Day 0 and a ≥ 4-fold increase in titer [1/dil] at Day 28
Number of participants with HAI antibody titer ≥ 40 [1/dil] against influenza H3 antigens | From Day 0 to Day 90
2-fold and 4-fold increase in SN antibody titers against influenza H3 antigens | From Day 0 to Day 90

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi Pasteur, a Sanofi Company
Locations (3):
- United States (3):
  - Research Centers of America Site Number : 8400002, Hollywood, Florida
  - Rochester Clinical Research, Inc. Site Number : 8400001, Rochester, New York
  - Coastal Carolina Research Center Site Number : 8400003, North Charleston, South Carolina

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: FBP00001 Plain Language Results Summary — https://sanofi.trialsummaries.com/Study/StudyDetails?id=25265&tenant=MT_SNY_9011